CLINICAL TRIAL: NCT01239329
Title: Understanding of Malnutrition in People With Complex Multiple Disabilities
Brief Title: Malnutrition in People With Complex Multiple Disabilities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Stichting Pergamijn (Gouverneur Kremers Centrum/azM) (Unknown); Koraalgroep(Gouverneur Kremers Centrum/azM) (Unknown); Lunetzorg (Gouverneur Kremers Centrum/azM) (Unknown)
Responsible Party: Prof. dr. L.M.G. Curfs, Maastricht University Medical Center
Other Study IDs: NL32655.068.10; MEC 10-2-043 (Other: Medical Ethical Committee University Hospital Maastricht)
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Complex Multiple Disabilities; Malnutrition
Keywords: Complex multiple disabilities; Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood as well as urine samples will be collected. Urine samples are important concerning measurement of body composition according to the Deuterium dilution method. A blood sample will be collected for measurement of nutrients.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Complex multiple disabilities: People with complex multiple disabilities, living in a care institution participating in the Governor Kremers Centre (GKC.)

SUMMARY:
Underweight is more prevalent in people with a mental handicap than in people without a mental handicap, especially in people with a severe mental handicap. It is unknown if these people are malnourished. There is no validated screening instrument available to determine the nutrition status in people with complex multiple disabilities. Research regarding malnutrition based on body composition and nutrients in stead of anthropometric data is important.

The aim of the study is to understand the nutritional status of people with complex multiple disabilitiest through measurement of body composition and nutritients. The primary objective of the study is: What percentage of people with complex multiple disabilities are malnourished, based on altered body composition and nutritients? Understanding the nutritional status of these patients is important in order for them to receive appropriate and effective treatment. This treatment is of interest for general health and the quality of daily life.

ELIGIBILITY:
Inclusion Criteria:

* Person with complex multiple disabilities;
* Living in a care institution participating in the Governor Kremers Centre (GKC);
* Chronically confined to a wheelchair or bedridden;
* 18+ years

Exclusion Criteria:

* Parenteral nutrition;
* Serious infection;
* Terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 125 people with complex multiple disabilities, living in a care institution participating in the Governor Kremers Centre (GKC).
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
What percentage of people with complex multiple disabilities are malnourished, based on altered body composition and nutritients? | One hour
  Concerning measurement of body composition, the Deuterium dilution method will be used. A blood sample will be collected for measurement of nutrients. Furthermore, clinical parameters (weight, height and abdominal girth) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Leopold MG Curfs, Professor, Study Director — Maastricht University Medical Center; Eric EJ Smeets, MD, Study Director — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands